CLINICAL TRIAL: NCT01632007
Title: Double-blind Comparative Study of SYR-472
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-472/CCT-002; U1111-1128-6104 (Registry Identifier: WHO); JapicCTI-121839 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — trelagliptin; alogliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SYR-472 100 mg (Experimental)
  Interventions: Drug: SYR-472
- Alogliptin 25 mg (Active Comparator)
  Interventions: Drug: Alogliptin 25 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYR-472
  Arms: SYR-472 100 mg
Drug: Alogliptin 25 mg
  Other Names: SYR-322
  Arms: Alogliptin 25 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of treatment with SYR-472 in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is an outpatient.
2. The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. The participant has any serious cardiac disease, serious cerebrovascular disorder, or any serious pancreatic or hematological disease.（e.g., subjects who require hospitalization or subjects who were hospitalized within 24 weeks prior to the commencement of the observation period)
2. The participant is considered ineligible for the study for any other reason by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2012-05-01 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2013-07-01 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) | 24 weeks.
  Measurement of change in HbA1c (ratio of hemoglobin bound to glucose).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda (Note: This product was divested to Teijin Pharma Limited in 2023)
Locations (22):
- Japan (22):
  - Akita, Akita
  - Matsudo-shi, Chiba
  - Fukuoka, Fukuoka
  - Fukuyama-shi, Hiroshima
  - Ishikari-shi, Hokkaido
  - Nakagawa-gun, Hokkaido
  - Sapporo, Hokkaido
  - Naka, Ibaragi
  - Sagamihara-shi, Kanagawa
  - Kumamoto, Kumamoto
  - Kashiwara-shi, Osaka
  - Osaka, Osaka
  - Suita-shi, Osaka
  - Arakawa-ku, Tokyo
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Katsushika-ku, Tokyo
  - Mitaka-shi, Tokyo
  - Shinjuku-ku, Tokyo
  - Shunan-shi, Yamaguchi

REFERENCES:
- [Derived] Inagaki N, Onouchi H, Maezawa H, Kuroda S, Kaku K. Once-weekly trelagliptin versus daily alogliptin in Japanese patients with type 2 diabetes: a randomised, double-blind, phase 3, non-inferiority study. Lancet Diabetes Endocrinol. 2015 Mar;3(3):191-7. doi: 10.1016/S2213-8587(14)70251-7. Epub 2015 Jan 19. PMID 25609193